#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for GSK2831781 study 207823: A randomised, double-blind, placebo-controlled Phase I study of the safety and tolerability, pharmacokinetics, and pharmacodynamics of a single intravenous dose of GSK2831781 in healthy Japanese and Caucasian participants, and a single subcutaneous dose of GSK2831781 in healthy Caucasian participants. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2831781 |
| Effective Date | : | 01-OCT-2019 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2018N393275\_01 of study 207823.
- This RAP is intended to describe the safety, tolerability, pharmacokinetics and pharmacodynamics analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analysis (IA) and Statistical Analysis Complete (SAC) deliverables.

# **RAP Author(s):**

| Approver | | Date | Approval Method |
|----------------|----------------|-------------|-----------------|
| Lead<br>PPD | | 27-SEP-2019 | Email |
| Statistician ( | Biostatistics) | | |
| Co-author | | 27-SEP-2019 | Email |
| Director (CP | MS) | 27-SE1-2019 | Eman |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmation:**

| Reviewer | Date | Confirmation<br>Method |
|---|---|---|
| Programming Manager (Biostatistics) | 26-SEP-2019 | Email |
| Physician Director, Discovery Medicine (CPEM) | 26-SEP-2019 | Email |

# **Other RAP Team Members:**

| Reviewer | Date | Confirmation<br>Method |
|--------------------------------------------|------|------------------------|
| Global Clinical Development Manager (GCSD) | N/A | N/A |
| Principal Clinical Data Manager (GCDO) | N/A | N/A |
| Director (SMG) | N/A | N/A |
| Group Leader (BIB-Immunogenicity) | N/A | N/A |
| Immunologist (Discovery Medicine) | N/A | N/A |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|-------------------------------------|-------------|--------------------------|
| Statistics Director (Biostatistics) | 30-SEP-2019 | Pharma TMF<br>eSignature |
| Programming Manager (Biostatistics) | 01-OCT-2019 | Pharma TMF<br>eSignature |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 6 |
| 2. | STIMM | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | |
| | | Changes to the Protocol Defined Statistical Analysis Plan | 0 |
| | 2.2. | Study Objectives and Endpoints | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Analyses | 10 |
| 3. | PLANI | NED ANALYSES | 11 |
| | 3.1. | Interim Analyses | 11 |
| | 3.2. | Final Analyses | |
| 4. | ΔΝΔΙ | YSIS POPULATIONS | 12 |
| \lnot. | 4.1. | Protocol Deviations | |
| | 4.1. | FIOLOGOI Deviations | 12 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 4.0 |
| | | /ENTIONS | |
| | 5.1. | General | |
| | 5.2. | Study Treatment & Sub-group Display Descriptors | |
| | 5.3. | Baseline Definitions | |
| | 5.4. | Examination of Strata | 14 |
| | 5.5. | Other Considerations for Data Analyses and Data Handling Conventions | 1/ |
| 6. | STUD | Y POPULATION ANALYSES | 15 |
| 7. | EFFIC | CACY ANALYSES | 16 |
| 8. | SAFE | TY ANALYSES | 17 |
| • | 8.1. | Adverse Events Analyses | |
| | 8.2. | Clinical Laboratory Analyses | |
| | 8.3. | Other Safety Analyses | |
| | 0.0. | Other Galety Analyses | 10 |
| 9. | | MACOKINETIC ANALYSES | |
| | 9.1. | Endpoint / Variables | |
| | | 9.1.1. Drug Concentration Measures | |
| | | 9.1.2. Derived Pharmacokinetic Parameters | 19 |
| | 9.2. | Summary Measure | 19 |
| | 9.3. | Population of Interest | |
| | 9.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 9.5. | Statistical Analyses / Methods | |
| | | 9.5.1. Statistical Methodology Specification (Part A) | |
| | | 9.5.2. Statistical Methodology Specification (Part B) | |
| 10 | P∪DII | JLATION PHARMACOKINETIC (POPPK) ANALYSES | ງງ |
| 10. | 10.1. | · | |
| | 10.1. | Statistical Arialyses / Interious | 22 |
| 11 | РНΔР | MACODYNAMIC ANALYSES | 23 |

| | 11.1. | Secondary Pharmacodynamic Analyses | |
|---|---|---|---|
| | | 11.1.1. Endpoint / Variables | |
| | | 11.1.2. Summary Measure | |
| | | 11.1.3. Population of Interest | |
| | | 11.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 11.1.5. Statistical Analyses / Methods | |
| | 11.2. | | |
| | | 11.2.1. Endpoint / Variables | |
| | | 11.2.2. Summary Measure | |
| | | 11.2.3. Population of Interest | |
| | | 11.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 11.2.5. Statistical Analyses / Methods | 24 |
| 12. | | RMACOKINETIC / PHARMACODYNAMIC ANALYSES | |
| | 12.1. | Statistical Analyses / Methods | 25 |
| 13. | | NOGENICITY ANALYSES | |
| | 13.1. | · · | |
| | 13.2. | Summary Measure | |
| | 13.3. | Population of Interest | |
| | 13.4. | · | |
| | 13.5. | Statistical Analyses / Methods | 26 |
| 14. | REFE | RENCES | 27 |
| 15. | | NDICES | |
| | 15.1. | 1.1 | |
| | 15.2. | 1 1 | |
| | | 15.2.1. Part A: Japanese and Caucasian Participants – IV dose | |
| | | 15.2.2. Part B: Caucasian Participants – SC dose | |
| | 15.3. | , , , | |
| | | 15.3.1. Definitions of Assessment Windows for Analyses | 36 |
| | 15.4. | Appendix 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | |
| | | 15.4.1. Study Phases for Parts A and B | |
| | | 15.4.1.1. Study Phases for Concomitant Medication | |
| | | 15.4.2. Treatment Emergent Flag for Adverse Events | |
| | 15.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | | 15.5.1. Reporting Process | |
| | | 15.5.2. Reporting Standards | |
| | | 15.5.3. Reporting Standards for Pharmacokinetic | |
| | 15.6. | Appendix 6: Derived and Transformed Data | |
| | | 15.6.1. General (Parts A and B) | |
| | | 15.6.2. Study Population | |
| | | 15.6.3. Safety | |
| | 15.7. | Appendix 7: Reporting Standards for Missing Data | |
| | | 15.7.1. Premature Withdrawals | |
| | | 15.7.2. Handling of Missing Data | |
| | | 15.7.2.1. Handling of Missing and Partial Dates | |
| | 15.8. | Appendix 8: Values of Potential Clinical Importance | |
| | | 15.8.1. Laboratory Values | |
| | | 15.8.2. ECG | 46 |

| | 15.8.3. | Vital Signs | 46 |
|--------|----------|-------------------------------------------------|----|
| | 15.8.4. | <b>-</b> | |
| 15.9. | Appendix | (9: Population Pharmacokinetic (PopPK) Analyses | 47 |
| | 15.9.1. | Population Pharmacokinetic (PopPK) Dataset | |
| | | Specification | 47 |
| | 15.9.2. | Population Pharmacokinetic (PopPK) Methodology | 47 |
| 15.10. | | (10: Pharmacokinetic / Pharmacodynamic Analyses | 48 |
| | 15.10.1. | Pharmacokinetic / Pharmacodynamic Dataset | |
| | | Specification | |
| | | Pharmacokinetic / Pharmacodynamic Methodology | |
| 15.11. | | 11: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 15.12. | | c 12: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | Pharmacokinetic Population (PopPK) Tables | |
| | | .Pharmacokinetic Population (PopPK) Figures | |
| | | .Pharmacodynamic Tables | |
| | | .Pharmacodynamic Figures | |
| | | .Pharmacokinetic / Pharmacodynamic Tables | |
| | | Pharmacokinetic / Pharmacodynamic Figures | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 15.13. | Appendix | (13: Example Mock Shells for Data Displays | 80 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|----------------------|-------------|-------------|
| 2018N393275_01 | 06-MAY-2019 | Amendment 1 |
| 2018N393275_00 | 13-MAR-2019 | Original |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Section 7.3 of the Protocol: a single Treatment Group B is defined for the active 150 mg SC dose. | Section 2.3 and Section 5.2 of the RAP: the active 150 mg SC dose in Part B corresponds to 3 treatment groups, coded B1, B2 and B3. | As described in the RCCS document, the randomised allocation of active dose to syringe 1, 2 or 3 is performed as part of the main randomisation effort. |

# 2.2. Study Objectives and Endpoints

| Objectives | | | Endpoints |
|---|---|---|---|
| Prim | nary | | |
| • | To evaluate the safety and tolerability after single IV dosing of GSK2831781 in healthy Japanese and Caucasian participants, and SC dosing in healthy Caucasian participants | • | AEs, vital signs, clinical laboratory values (haematology, clinical chemistry, and urinalysis), 12-lead ECG Local tolerability |
| Seco | ondary | | |
| • | To evaluate the PK of GSK2831781 after a single IV dose in healthy Japanese and Caucasian participants (Part A) | • | GSK2831781 PK parameters following single IV dose: area under the plasma concentration-time curve [AUC(0-t)], maximum observed plasma concentration (Cmax), time of occurrence of Cmax (tmax) |
| • | To evaluate the PK of GSK2831781 after a single SC dose in healthy Caucasian participants (Part B) | • | GSK2831781 PK parameters following single SC dose: AUC(0-t), Cmax, tmax, bioavailability (F) |

| | Objectives | | Endpoints |
|---|---|---|---|
| • | To evaluate the effect of a single IV or SC dose of GSK2831781 on depletion of LAG3+T cells in blood | | PK/PD relationship between plasma PK of GSK2831781 and LAG3+ T cells in blood over time |
| • | To investigate the immunogenicity of single IV and SC doses of GSK2831781 | • | ADAs over time |
| Exp | loratory | | |
| • | To evaluate the concentration-time profiles of GSK2831781 after a single IV dose in healthy Japanese and Caucasian participants (Part A) | | GSK2831781 PK concentrations over time following single IV dose |
| • | To evaluate the concentration-time profiles of GSK2831781 after a single SC dose in healthy Caucasian participants (Part B) | | GSK2831781 PK concentrations over time following single SC dose |
| • | To evaluate the effect of a single IV or SC dose of GSK2831781 on soluble LAG3 (sLAG3) concentrations | | Soluble LAG3 (sLAG3) concentrations in blood over time |
| • | To evaluate the effect of GSK2831781 on regulatory T cells in blood | | PK/PD relationship between plasma PK of GSK2831781 and regulatory T cells in blood over time |

# 2.3. Study Design

This study is a double-blind, placebo-controlled, randomised, parallel group, two-part study, with single IV doses administered to healthy Japanese and Caucasian participants, or SC doses administered to healthy Caucasian participants.

In Part A, single IV doses of 450 mg GSK2831781 or placebo will be administered to Japanese or Caucasian healthy participants, with stratification by ethnicity.

In Part B, single SC doses of 150 mg or 450 mg GSK2831781, or placebo, will be administered to healthy Caucasian participants.

At least one interim analysis will be conducted during the study (see Section 3.1 for further details).

In line with routine pharmacovigilance, an internal GSK Safety Review Team (SRT) (which will include a subset of the 207823 study team) will review blinded safety data, including clinical laboratory parameters and adverse events, at appropriate intervals during the period of study conduct.



| Part A: Overview of | of Study Design and | Key Features |
|---|---|---|
| Part A Design<br>Features | <ul> <li>Part A will be a single centre, parallel group, single dose part. It is designed to investigate whether there are any differences due to ethnicity in safety and tolerability, or PK and PK/PD relationship in blood between healthy Japanese and Caucasian participants following a single IV 450 mg dose of GSK2831781.</li> <li>Separate cohorts of participants will be enrolled into Parts A and B.</li> <li>Part A will consist of a single cohort of 16 healthy participants, stratified by ethnicity: 8 participants will be Japanese and 8 will be Caucasian. Up to a maximum of 32 participants may be enrolled if a dose reduction is needed.</li> <li>The participants in each ethnicity stratum will be randomised in a 3:1 ratio to receive either 450 mg GSK2831781 IV or placebo. If a dose reduction is needed, the new participants in each ethnicity stratum will also be randomised in a 3:1 ratio to receive either GSK2831781 IV or placebo.</li> <li>Part A study duration, including screening and follow-up, is not expected to exceed 147 days for any participant.</li> </ul> | |
| Part A Dosing | <ul> <li>Participants will be dosed once on day 1.</li> <li>In Part A, in order to bridge from the first-time-in human study (GSK Study 200630), dosing episodes will initially be separated by a minimum of 22 hours, until 3 participants in one of the strata have been dosed and monitored for a minimum of 46 hours. Subsequently, the remaining participants in Part A will be dosed, unless stopping criteria have been met.</li> </ul> | |
| Part A Time & Events | Refer to Appendix 2. | |
| Part A<br>Treatment<br>Assignment | Participants will be assigned to either 450mg GSK2831781 IV or placebo in a 3:1 ratio, stratified by ethnicity. The treatment codes will be: | |
| | Treatment code Treatment Description | |
| | A 450 mg GSK2831781 IV | |
| | Р | P Placebo IV |

| Part A: Overview | Part A: Overview of Study Design and Key Features |
|---|---|
| | If a dose reduction is needed, the new participants in each ethnicity stratum will also be randomised in a 3:1 ratio to receive either GSK2831781 IV or placebo, according to the randomisation schedule. |
| Part A Interim<br>Analysis | <ul> <li>An interim analysis for Part A will be performed once at least 8 participants in each stratum have completed their Day 8 visit, and at least 6 participants in each stratum have completed their Day 29 visit, where Safety, PK and PD data will be reviewed.</li> <li>See Section 3.1 for further details.</li> </ul> |

| Part B: Overview of | of Study Design and Ke | y Features |
|---|---|---|
| Part B: Overview of Part B Design Features | <ul> <li>Once the final Caurecruitment to Part</li> <li>Part B will be a single explore the safety a single dose of SC (healthy Caucasian)</li> <li>As the 450 mg dos participants randon injections (using 0.5 maintain the blind. one of the three systems of the systems of the systems of the participants with GSK2831781 SC, 4</li> <li>The 8 planned 150 3 in a 3:3:2 ratio.</li> </ul> | final Caucasian participant is recruited into Part A of the study, nt to Part B may commence. Il be a single centre, parallel group, single dose part. It is designed to be safety and tolerability, PK and PK/PD relationship in blood following a see of SC GSK2831781 at 150 mg and 450 mg dose levels, or placebo, in saucasian participants. If one dose level requires 3 injections of GSK2831781 150 mg, and the standomised to the 150 mg dose level or placebo will also receive 3 (using 0.9% saline placebo as dummy injections, where needed) to the blind. In the 150 mg case, the allocation of active GSK2831781 to be three syringes will be randomised. If consist of participants will be enrolled into Parts A and B. If consist of a single cohort of 20 healthy Caucasian participants. Up to a performance of 30 participants may be enrolled if a dose reduction is needed. Scipants will be randomised in a 2:2:1 ratio to receive 150 mg and 150 mg participants will be randomly allocated active syringe 1, 2 or 2:2 ratio. |
| Part B Dosing | <ul><li>Participants will be</li><li>In Part B, as this w<br/>sentinel dosing will</li></ul> | |
| Part B Time & Events | Refer to Appendix | • |
| Part B<br>Treatment<br>Assignment | Participants will be assigned to 150 mg GSK2831781 SC or 450 mg GSK2831781 SC or placebo in a 2:2:1 ratio. The treatment codes will be: | |
| | Treatment code Tr | Treatment code Treatment Description |
| | B1 150 mg GSK2831781 SC injection 1 active | |
| | B2 15 | B2 150 mg GSK2831781 SC injection 2 active |
| | B3 15 | 50 mg GSK2831781 SC injection 3 active |

| Part B: Overview of Study Design and Key Features | | |
|---|---|---|
| | С | 450 mg GSK2831781 SC |
| Q | | Placebo SC |
| Part B Interim<br>Analysis | No interim and | No interim analyses will be performed during Part B. |

# 2.4. Statistical Analyses

The primary objective of this study is to determine the safety and tolerability of a single intravenous dose of GSK2831781 in healthy Japanese and Caucasian participants, and a single subcutaneous dose of GSK2831781 in healthy Caucasian participants. No formal hypotheses will be tested.

An estimation approach will be used to describe pharmacokinetics of GSK2831781, where point estimates and corresponding 90% confidence intervals will be constructed, unless otherwise stated.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis for Part A will be performed once at least 8 participants in each stratum have completed their Day 8 visit, and at least 6 participants in each stratum have completed their Day 29 visit, where Safety, PK and PD data will be reviewed. The interim analysis will be utilised to determine if Japanese participants can be recruited into the Phase 2 study (204869) under the existing dosing strategy.

An Interim Data Review Committee (DRC) will be utilised in this study to review the interim analysis data. The DRC will be composed of a limited number of people, who may be members of the 207823 study team, including the statistician, a senior safety representative, lead physician and the pharmacokineticist. A DRC Charter will contain the details regarding the DRC, including membership, decision rules for the interim, and required data integrity and data quality control.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in Section 5.4 of the protocol: the end of the study is defined as the date of the last visit (including follow-up) of the last participant in the study (Parts A and B).
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) have been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Description | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility. | Study Population<br>(specific only) |
| Randomized | All participants who are randomised into the study and receive a randomisation number. | Study Population<br>(specific only) |
| Safety | All Randomized participants who receive study intervention. Participants will be analysed according to the intervention they actually received. | <ul><li>Study Population</li><li>Safety</li><li>PD</li><li>PK/PD</li></ul> |
| Pharmacokinetic (PK) | All Safety participants for whom a PK sample was obtained and analysed. Participants will be analysed according to the intervention they actually received. | • PK |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

Note that a participant is considered evaluable if they have been dosed and have safety and PK data up to Day 29 (Parts A and B).

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This output will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

#### 5.1. General

Parts A and B will be reported separately, with separate outputs generated for each, unless stated otherwise.

# 5.2. Study Treatment & Sub-group Display Descriptors

In the Tables, Listings and Figures (TLF), treatment should be presented with placebo first, then in order of increasing dose within each part.

| Part A: Treatment Groups Descriptions | | | |
|---|---|---|---|
| | Randall NG Data Displays for Reporting | | |
| Code | Description | Order in TLF | |
| Α | 450 mg GSK2831781 IV | 450 mg GSK2831781 IV | 2 |
| Р | Placebo IV | Placebo IV | 1 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. 450 mg GSK2831781 IV vs Placebo IV

A subset of Part A data displays will be presented with a combination of treatment groups and geographic ancestry stratification, as described in Section 5.4.

| Part B: Treatment Groups Descriptions | | | |
|---|---|---|---|
| | Randall NG Data Displays for Reporting | | |
| Code | Code Description Description | | |
| B1 | 150 mg GSK2831781 SC injection 1 active | 150 mg GSK2831781 SC injection<br>1 | 2 (*) |
| B2 | 150 mg GSK2831781 SC injection 2 active | 150 mg GSK2831781 SC injection 2 | 3 (*) |
| B3 | 150 mg GSK2831781 SC injection 3 active | 150 mg GSK2831781 SC injection 3 | 4 (*) |
| С | 450 mg GSK2831781 SC | 450 mg GSK2831781 SC | 5 |
| Q | Placebo SC | Placebo SC | 1 |

(\*) Note that treatment groups B1, B2 and B3 will be combined into a single "150 mg GSK2831781 SC" group in most tables, figures and listings. Only a small subset of outputs, including listings of injection site reactions (Section 15.12 for details), will report B1, B2 and B3 as separate treatment groups.

Treatment comparisons will be displayed as follows using the descriptors as specified, where "150 mg GSK2831781 SC" includes treatment groups B1, B2 and B3:

- 1. 150 mg GSK2831781 SC vs Placebo SC
- 2. 450 mg GSK2831781 SC vs Placebo SC

#### 5.3. Baseline Definitions

- The baseline value (in both Parts A and B) will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
- If time is not collected, Day 1 assessments are assumed to be taken prior to dosing and used as baseline.
- Replicate assessments at a timepoint will be averaged, and the mean value will be used.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.4. Examination of Strata

The list of strata may be used in descriptive summaries and statistical analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | Part A: stratification by geographic ancestry (Caucasian vs Japanese). |
| | Used for ethnosensitivity comparisons. |
| | A subset of Part A data displays will be presented with the following groups, in this |
| | order: |
| | <ul> <li>Placebo (Caucasian)</li> </ul> |
| | <ul> <li>Placebo (Japanese)</li> </ul> |
| | <ul> <li>450 mg GSK2831781 (Caucasian)</li> </ul> |
| | <ul> <li>450 mg GSK2831781 (Japanese)</li> </ul> |

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 15.3 | Appendix 3: Assessment Windows |
| 15.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 15.6 | Appendix 6: Derived and Transformed Data |
| 15.7 | Appendix 7: Reporting Standards for Missing Data |
| 15.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Details of the planned displays are presented in Appendix 12: List of Data Displays.

# 7. EFFICACY ANALYSES

There are no efficacy analyses to be included in this study.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 8.1. Adverse Events Analyses

The definition of an AE is detailed in Appendix 3 of the protocol.

Analyses of AEs will include those events that are Treatment Emergent as defined in Section 15.4.

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and Liver function tests will be based on GSK Core Data Standards.

Clinical laboratory summaries will include all assessments post-baseline. All clinical laboratory assessments, including pre-baseline (i.e. screening), will be listed.

The details of the planned displays are in Appendix 12: List of Data Displays.

The laboratory assessments for each category are displayed below (Table 1 in Section 11.2 of the protocol):

| Laboratory<br>Assessments | Parameters | | | | | |
|---|---|---|---|---|---|---|
| Haematology | Platelet Count Red Blood Cell (RBC) Count Haemoglobin Haematocrit | | RBC Indices: Mean Corpuscular Volume (MCV) Mean Corpuscular Haemoglobin (MCH) %Reticulocytes | | White Blood Cell (WBC) count with Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils | |
| Clinical<br>Chemistry <sup>1</sup> | Blood Urea<br>Nitrogen (BUN) | Potas | sium | Aspartate Aminotransfer (AST)/Serum Glutamic- Oxaloacetic Transaminase (SGOT) | | Total and direct bilirubin |
| | Creatinine Estimated Glomerular Filtration Rate (eGFR) | Sodium | | Alanine<br>Aminotransfer<br>(ALT/Serum<br>Glutamic-Pyru<br>Transaminase | vic | Total Protein |

| Laboratory<br>Assessments | Parameters | | | |
|---|---|---|---|---|
| | (SGPT) | | | |
| | Glucose [non-<br>fasting] | Calcium | Alkaline phosphatase | |
| Routine<br>Urinalysis | Specific gravity | | | |
| · | <ul> <li>pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> | | | |
| Other Screening<br>Tests (not to be<br>reported) | opiates, cannab | en (to include at minin<br>inoids and benzodiaz | , | |
| | <ul> <li>Serology: HIV a<br/>antibody<sup>3</sup>, VZV</li> </ul> | | .b, HCV antibody, EBV a | ntibody <sup>3</sup> , CMV |
| | Quantiferon test | t for TB | | |

#### NOTES:

- 1. Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are given in Section 8.2.3 of the protocol. All events of ALT ≥3 × upper limit of normal (ULN) and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).
- 2. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.
- 3. To be repeated in event of possible viral reactivation.

Laboratory results that could unblind the study will not be reported to investigative sites or other blinded personnel until the study has been unblinded.

# 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

The non-laboratory safety test results include:

- ECGs
- Vital signs
- Local tolerability

The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 9. PHARMACOKINETIC ANALYSES

# 9.1. Endpoint / Variables

# 9.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 15.5.3 Reporting Standards for Pharmacokinetic).

#### 9.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times.

Pharmacokinetic parameters listed will be determined from the plasma concentrationtime data, as data permits. Additional parameters may be included as required.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of last quantifiable concentration (C(t)). |
| | Calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration. |
| | Determined directly from the concentration-time data. |
| tmax | Time to reach Cmax. |
| | Determined directly from the concentration-time data. |

# 9.2. Summary Measure

Descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum) will be calculated by treatment (and geographic ancestry in Part A) for all PK concentrations over time and for the derived PK parameters. In addition, for log-transformed PK parameter variables, geometric mean, 95% CI and %CV<sub>b</sub> will be provided.

# 9.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 9.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

• Withdrawn participants may be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant.

- All available data from participants who were withdrawn from the study will be analysed and listed, and all available planned data will be included in summary tables and figures, unless otherwise specified.
- Missing and anomalous concentration data not due to intercurrent events will be handled according to SOP 314000.

# 9.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 9.5.1. Statistical Methodology Specification (Part A)

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma concentration-time profiles).

#### **Ethnosensitivity (Part A)**

#### **Endpoint / Variables**

- AUC(0-t)
- Cmax

#### Model Specification

- Analysis of variance (ANOVA) will be performed on log-transformed data to determine the point estimate for the comparison of Japanese to Caucasian participants.
- This analysis will be repeated for each of the PK parameters at the 450 mg dose level.
- The 90% confidence interval for the mean difference of the log-transformed data will be calculated. The equivalent 90% confidence interval for the geometric means will be provided.

#### **Model Checking & Diagnostics**

- Normality assumptions underlying the model used for analysis will be examined by obtaining a normal
  probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the
  normality assumption and constant variance assumption of the model, respectively) to gain confidence
  that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- Table of:
  - Geometric means and ratio of geometric means with 90% CI.

#### 9.5.2. Statistical Methodology Specification (Part B)

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma concentration-time profiles).

Note that the intravenous PK data for bioavailability analyses will be taken from the Caucasian stratum in Part A.

#### **Bioavailability (Part B)**

#### **Endpoint / Variables**

AUC(0-t)

#### **Model Specification**

- Analysis of variance (ANOVA) will be performed on log-transformed data to determine the point estimate for the comparison of SC and IV administration.
- The resulting estimated difference is the log point estimate of the absolute bioavailability (Fabs).
- This analysis will be conducted at the 450 mg dose level only.
- The 90% confidence interval for the mean difference of the log-transformed data will be calculated. The equivalent 90% confidence interval for the geometric means will be provided.

#### **Model Checking & Diagnostics**

- Normality assumptions underlying the model used for analysis will be examined by obtaining a normal
  probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the
  normality assumption and constant variance assumption of the model, respectively) to gain confidence
  that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- Table of:
  - o Geometric means and ratio of geometric means with 90% Cl.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

The primary goal of this analysis is to characterize the population pharmacokinetics of GSK2831781 administered IV in Japanese and Caucasian healthy volunteers and SC in Caucasian healthy volunteers. The individual participant PK parameters will be estimated and documented for the purposes of any subsequent exposure-response (PK/PD) analyses. Any inter-ethnic differences in the PK will also be investigated.

# 10.1. Statistical Analyses / Methods

A summary of the planned population pharmacokinetic analyses is outlined below:

- A previous PopPK model developed based on the drug plasma and total serum sLAG3 concentrations collected during the first-time in human study 200630 (GSK Document Number 2017N352860\_00) will be fitted to the drug plasma concentration-time data using the nonlinear mixed effects modelling software NONMEM.
- Individual post-hoc estimated PK parameters will be summarised descriptively.
- To support this analysis a PopPK dataset will be generated. The details for the dataset specifications are provided in Appendix 9: Population Pharmacokinetic (PopPK) Analyses.

Detailed PopPK methodology is presented in Appendix 9: Population Pharmacokinetic (PopPK) Analyses.

#### 11. PHARMACODYNAMIC ANALYSES

# 11.1. Secondary Pharmacodynamic Analyses

#### 11.1.1. Endpoint / Variables

| Parameter | Parameter Description |
|---|---|
| LAG3+ | <ul> <li>LAG3+ T cell numbers and frequencies in blood. The following cell populations will be<br/>reported:</li> </ul> |
| | ○ CD4+CD45RA-J11L1+ |
| | ○ CD4+CD45RA-REA351+ |
| | ○ CD4 <sup>-</sup> CD45RA <sup>-</sup> J11L1 <sup>+</sup> |
| | ○ CD4-CD45RA-REA351+ |

# 11.1.2. Summary Measure

Absolute value and percent change from baseline (%CFB) are of interest.

Part A: Data will be available at baseline and at day 1 (6h, 24h), 4, 8, 15, 29, 43, 57, 85 and 112.

Part B: Data will be available at baseline and at day 2, 4, 8, 15, 29, 43, 57, 85 and 112.

#### 11.1.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the Safety population, unless otherwise specified.

#### 11.1.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

- Withdrawn participants may be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant.
- All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.

#### 11.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 11.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

## 11.2. Exploratory Pharmacodynamic Analyses

#### 11.2.1. Endpoint / Variables

| Parameter | Parameter Description |
|---|---|
| sLAG3 | Concentration of soluble LAG3 in blood. |
| Regulatory T cells | CD3+CD4+CD45RA-CD25+CD127 <sup>Io</sup> FoxP3+ Regulatory T cell numbers and frequencies in blood |

#### 11.2.2. Summary Measure

Absolute value and percent change from baseline (%CFB) are of interest.

#### sLAG3:

Part A: Data will be available at baseline and at day 1 (1h, 2h, 6h, 12h, 24h), 3, 4, 8, 15, 22, 29, 43, 57, 71, 85 and 112.

Part B: Data will be available at baseline and at day 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 112.

#### **Regulatory T cells:**

Part A: Data will be available at baseline and at day 4 and 112.

#### 11.2.3. Population of Interest

The exploratory pharmacodynamics analyses will be based on the Safety population, unless otherwise specified.

#### 11.2.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

- Withdrawn participants may be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant.
- All available data from participants who were withdrawn from the study will be listed
  and all available planned data will be included in summary tables and figures, unless
  otherwise specified.

# 11.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 11.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The primary goal of this analysis is to characterize the pharmacokinetic / pharmacodynamic (PK/PD) relationship of GSK2831781 administered IV in Japanese and Caucasian healthy volunteers and SC in Caucasian healthy volunteers. Any interethnic differences in the PK/PD relationship will also be investigated.

# 12.1. Statistical Analyses / Methods

A summary of the planned population PK/PD analyses are outlined below:

- A previous PopPK/PD model developed based on the individual post hoc predicted PK parameters and all available cell depletion data from the first-time in human study 200630 (GSK Document Number 2017N352860\_00) will be fitted to the drug plasma concentration (or PK parameters) and PD data using the nonlinear mixed effects modelling software NONMEM.
- To support this analysis a PK/PD dataset will be generated. The details for the dataset specifications are provided in Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses.
- Detailed PK/PD methodology is presented in Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses.

#### 13. IMMUNOGENICITY ANALYSES

#### 13.1. Endpoint / Variables

| Parameter | Parameter Description |
|-----------|---------------------------------|
| ADAs | Anti-drug antibodies over time. |

# 13.2. Summary Measure

Incidence and duration of anti-drug antibodies (ADA).

The GSK2831781 immunogenicity response will be summarized for the binding antibody assay by treatment group and timepoint. The table will include the number and proportion of participants in each result category for each visit. Binding confirmatory assay results will be categorized as Negative, Positive, or Unknown. Positive samples in the binding assay are further categorized as Transient Positive (i.e. single positive response that does not occur at the final assessment) or Persistent Positive (i.e. positive response that occurs at least 2 consecutive assessments or a single result at the final assessment). Titre for samples confirming positive in the binding assay will be reported in listings.

Parts A and B: Data will be available at baseline and at day 29, 57, 85 and 112.

# 13.3. Population of Interest

The immunogenicity analyses will be based on the Safety population, unless otherwise specified.

# 13.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

- Withdrawn participants may be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant.
- All available data from participants who were withdrawn from the study will be listed
  and all available planned data will be included in summary tables and figures, unless
  otherwise specified.

# 13.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 13.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 14. REFERENCES

GSK Document Number 2018N393275\_01. Study ID 207823: A randomised, double-blind, placebo-controlled Phase I study of the safety and tolerability, pharmacokinetics, and pharmacodynamics of a single intravenous dose of GSK2831781 in healthy Japanese and Caucasian participants, and a single subcutaneous dose of GSK2831781 in healthy Caucasian participants. 06-MAY-2019.

GSK Document Number 2017N352860\_00. Study ID 200630: A randomised, double blind (sponsor unblinded), placebo controlled, single ascending dose study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a IV dose of GSK2831781 in healthy volunteers and patients with plaque psoriasis.

# 15. APPENDICES

# 15.1. Appendix 1: Protocol Deviation Management

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan. Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset. This dataset will be the basis for the summaries and listings of protocol deviations.

# 15.2. Appendix 2: Schedule of Activities

# 15.2.1. Part A: Japanese and Caucasian Participants – IV dose

| | Screeni<br>ng | | | | ] | Day 1 (Ho | urs) | | | | | | | Day | s 3 – 8 | 35 | | | | Follow<br>Up/Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (up to<br>28 days<br>before<br>Dosing) | Day -1 | Pre-<br>Dose | 0<br>h <sup>1</sup> | 1 h | 2 h<br>(end of<br>infusio<br>n) | 6 h | 12 h | 24 h | 3 2 | 4 2 | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 85 | Withdra<br>wal (112<br>Days<br>post<br>dose) <sup>3</sup> |
| Window | | | -60<br>min | | ±10<br>min | +30<br>min <sup>4</sup> | ±30<br>min | ±30<br>min | ±60<br>min | | | ±1<br>d | ±2<br>d | ±2<br>d | ±2<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±7d |
| Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | |
| Inclusion and Exclusion Criteria | X | X | | | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | | | | |
| Full physical examination including height and weight | X | | | | | | | | | | | | | | | | | | | X |
| Medical history<br>(includes<br>substance usage) | X | | | | | | | | | | | | | | | | | | | |
| Past and Current<br>Medical<br>Conditions | X | | | | | | | | | | | | | | | | | | | |

| | Screeni<br>ng<br>(up to | Da | | | ] | Day 1 (Hot | urs) | | | | | | | Day | rs 3 – 8 | 35 | | | | Follow<br>Up/Early<br>Withdra |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | 28 days<br>before<br>Dosing) | Day -1 | Pre-<br>Dose | 0<br>h <sup>1</sup> | 1 h | 2 h<br>(end of<br>infusio<br>n) | 6 h | 12 h | 24 h | 3 2 | 4 2 | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 85 | wal (112<br>Days<br>post<br>dose) <sup>3</sup> |
| Window | | | -60<br>min | | ±10<br>min | +30<br>min <sup>4</sup> | ±30<br>min | ±30<br>min | ±60<br>min | | | ±1<br>d | ±2<br>d | ±2<br>d | ±2<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±7d |
| Serology (HIV,<br>HBV, HCV,<br>CMV, EBV,<br>VZV) | X | | | | | | | | | | | | | | | | | | | |
| TB screening<br>(QuantiFERON<br>± PPD) | X | | | | | | | | | | | | | | | | | | | |
| Breath Alcohol<br>Screen | X | X | | | | | | | | | | | | | | | | | | |
| Urine Drug<br>Screen | X | X | | | | | | | | | | | | | | | | | | |
| Haematology & Clinical Chemistry | X | X | | | | | | | X | X | | X | X | | X | X | X | | X | X |
| Urinalysis | X | X | | | | | | | X | X | | X | X | | X | X | X | | X | X |
| 12-Lead ECG <sup>5</sup> | X | | X | | | | X | | X | | | | | | | | | | X | X |
| Vital Signs <sup>6</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| Procedure | Screeni<br>ng<br>(up to<br>28 days<br>before<br>Dosing) | Day -1 | Pre-<br>Dose | 0<br>h <sup>1</sup> | 1 h | Day 1 (Hou<br>2 h<br>(end of<br>infusio<br>n) | urs)<br>6 h | 12 h | 24 h | 3 2 | 4 2 | 8 | 15 | Day | 29 | 43 | 57 | 71 | 85 | Follow<br>Up/Early<br>Withdra<br>wal (112<br>Days<br>post<br>dose) <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Window | | | -60<br>min | | ±10<br>min | +30<br>min <sup>4</sup> | ±30<br>min | ±30<br>min | ±60<br>min | | | ±1<br>d | ±2<br>d | ±2<br>d | ±2<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±7d |
| Randomization | | X | | | | | | | | | | | | | | | | | | |
| IMP<br>Administration | | | | <=====> | | | | | | | | | | | | | | | | |
| Resident in unit | | | <===== | ==================================== | | | | | | | | | | | | | | | | |
| Local<br>Tolerability | | | X | | | X | X | X | X | | | | | | | | | | | |
| sLAG3 concentrations | | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PK | | | X | | X | $X^7$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Immunogenicity | | | X | | | | | | | | | | | | X | | X | | X | X |
| LAG3 <sup>+</sup> Cell<br>Depletion and<br>Immunophenoty<br>ping | | | X | | | | X | | X | | X | X | X | | X | X | X | | X | X |
| Genetic Sample <sup>8</sup> | | | X | | | | | | | | | | | | | | | | | |
| AE/ SAE<br>Review | | | SAEs | colle | cted from | signing of | informed | l consent | form; AE | s col | lecte | d con | tinuou | ısly fr | om tin | ne of | first d | ose. | | |
| Concomitant<br>Medication | | | | | M | Ionitored f | rom scree | ening unti | the end | of the | e fina | al trea | tment | perio | d. | | | | | |

| | Screeni<br>ng | | | | ĵ | Day 1 (Hou | ırs) | | | | | | | Day | rs 3 – 8 | 35 | | | | Follow<br>Up/Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (up to<br>28 days<br>before<br>Dosing) | Day -1 | Pre-<br>Dose | 0<br>h <sup>1</sup> | 1 h | 2 h<br>(end of<br>infusio<br>n) | 6 h | 12 h | 24 h | 3 2 | 4 2 | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 85 | Withdra<br>wal (112<br>Days<br>post<br>dose) <sup>3</sup> |
| Window | | | -60<br>min | | ±10<br>min | +30<br>min <sup>4</sup> | ±30<br>min | ±30<br>min | ±60<br>min | | | ±1<br>d | ±2<br>d | ±2<br>d | ±2<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±3<br>d | ±7d |
| Review | | | | | | | | | | - | | | | | | | | | | |

#### Footnotes:

- 1. All post dose time points are in reference to the start of infusion.
- 2. Assessments at these visits should be on the scheduled day however can be at any time in the day.
- 3. Early withdrawal assessments will be the same as Follow-Up.
- 4. End of infusion assessment time window is +30 minutes for all assessments except for the PK sample which should be collected just before the end of the infusion.
- 5. ECG in triplicate at screening and single at all other time points.
- 6. Vital Signs to be taken every 30 minutes from start of infusion until completion of 2hr post dose monitoring period.
- 7. PK sample at end of infusion should be collected just before the end of the infusion.
- 8. The genetic sample is optional and can be taken any time after consent has been signed and the participant is randomized.

# 15.2.2. Part B: Caucasian Participants – SC dose

| | | | Г | Day 1 | | | | | | | | Days | 2-85 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 28 days<br>before Dosing) | Day - 1 | Pre-Dose | 0h | Post Dose <sup>1</sup> | 22 | 32 | 42 | 62 | 8 | 11 | 15 | 18 | 22 | 29 | 43 | 57 | 71 | 85 | Follow Up/Early<br>Withdrawal (112<br>Days post dose) <sup>3</sup> |
| Window | | | -60<br>min | | | | | | | ±1d | ±2d | ±2d | ±2d | ±2d | ±2d | ±3d | ±3d | ±3d | ±3d | ±7d |
| Informed consent | X | | | | | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | X | X | | | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | | | | |
| Full physical examination including height and weight | X | | | | | | | | | | | | | | | | | | | X |
| Medical history<br>(includes substance<br>usage) | X | | | | | | | | | | | | | | | | | | | |
| Past and current medical conditions | X | | | | | | | | | | | | | | | | | | | |
| Serology (HIV,<br>HBV, HCV, CMV,<br>EBV, VZV) | X | | | | | | | | | | | | | | | | | | | |
| TB screening<br>(QuantiFERON ±<br>PPD) | X | | | | | | | | | | | | | | | | | | | |

| | | | Г | Day 1 | | | | | | | | Days | 2-85 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 28 days<br>before Dosing) | Day - 1 | Pre-Dose | 0h | Post Dose <sup>1</sup> | 22 | 32 | 42 | 62 | 8 | 11 | 15 | 18 | 22 | 29 | 43 | 57 | 71 | 85 | Follow Up/Early<br>Withdrawal (112<br>Days post dose) <sup>3</sup> |
| Window | | | -60<br>min | | | | | | | ±1d | ±2d | ±2d | ±2d | ±2d | ±2d | ±3d | ±3d | ±3d | ±3d | ±7d |
| Breath Alcohol<br>Screen | X | X | | | | | | | | | | | | | | | | | | |
| Urine Drug Screen | X | X | | | | | | | | | | | | | | | | | | |
| Haematology & Clinical Chemistry | X | X | | | | X | X | | | X | | X | | | X | X | X | | X | X |
| Urinalysis | X | X | | | | X | X | | | X | | X | | | X | X | X | | X | X |
| 12-Lead ECG <sup>4</sup> | X | | X | | X <sup>5</sup> | X | | | | | | | | | | | | | X | X |
| Vital Signs <sup>6</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization | | X | | | | | | | | | | | | | | | | | | |
| IMP Administration | | | | $X^7$ | | | | | | | | | | | | | | | | |
| Resident in Unit | | <= | | | | => | | | | | | | | | | | | | | |
| Local tolerability at injection sites | | | X | | X8 | X | | X | | X | | | | | | | | | | |
| sLAG3 concentrations | | | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PK | | | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Immunogenicity | | | X | | | | | | | | | | | | X | | X | | X | X |

| | | | Γ | Day 1 | | | | | | | | Days | 3 2-85 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 28 days<br>before Dosing) | Day - 1 | Pre-Dose | 0h | Post Dose <sup>1</sup> | 22 | 32 | 42 | 62 | 8 | 11 | 15 | 18 | 22 | 29 | 43 | 57 | 71 | 85 | Follow Up/Early<br>Withdrawal (112<br>Days post dose) <sup>3</sup> |
| Window | | | -60<br>min | | | | | | | ±1d | ±2d | ±2d | ±2d | ±2d | ±2d | ±3d | ±3d | ±3d | ±3d | ±7d |
| LAG3 <sup>+</sup> Cell<br>Depletion | | | X | | | X | | X | | X | | X | | | X | X | X | | X | X |
| Genetic Sample <sup>9</sup> | | | X | | | | | | | | | | | | | | | | | |
| AE/SAE Review | SAEs collected f | rom s | igning of | finfor | med c | onsen | t form | ; AEs | colle | cted c | ontin | uously | from | time | of firs | st dose | ). | | | |
| Concomitant medication review | Monitored from | scree | ning unti | l the e | end of | the fi | nal tre | atmer | nt peri | od. | | | | | | | | | | |

#### Footnotes:

- 1. All post dose time points are in reference to the first injection of IMP.
- 2. Assessments at these visits should be on the scheduled day however can be at any time in the day.
- 3. Early withdrawal assessments will be the same as Follow-Up.
- 4. ECG in triplicate at screening and single at all other time points.
- 5. ECG to be performed 6 hours post dose.
- 6. Vital Signs to be taken every 30 minutes from first IMP injection until completion of 2hr post dose monitoring period.
- 7. IMP administration consists of 3 syringes, all 3 syringes are to be administered as closely together as possible (preferably within 10 minutes).
- 8. Post dose Local tolerability at injection sites to be reviewed at 2, 6, 12, and 24 hours post dose.
- 9. The genetic sample is optional and can be taken any time after consent has been signed and the participant is randomized.

# 15.3. Appendix 3: Assessment Windows

# 15.3.1. Definitions of Assessment Windows for Analyses

No assessment windows will be defined for analyses. Summaries and analyses will be based on nominal visits.
# 15.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 15.4.1. Study Phases for Parts A and B

Assessments and events will be classified according to the time of occurrence relative to the dose.

| Study Phase | Definition |
|--------------------|---------------------------------------------|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| Treatment Emergent | Date/Time > Study Treatment Start Date/Time |

#### 15.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to study treatment. |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 15.4.2. Treatment Emergent Flag for Adverse Events

Adverse Events will be flagged as Treatment Emergent as described in the table in Section 15.4.1, where the AE Start Date/Time will be considered.

# 15.5. Appendix 5: Data Display Standards & Handling Conventions

## 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supply | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound | Each of the following directories will be used for both Parts A and B. : \arprod\gsk2831781\mid207823\internal_01 : \arprod\gsk2831781\mid207823\interim_01 : \arprod\gsk2831781\mid207823\final_01 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Integrated Data Standards Library (IDSL) GSK A&amp;R<br/>dataset standards.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be get a second control of the second control | enerated for SAC. |

#### 15.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

| Unscheduled visits | Unscheduled visits will not be included in summary tables and/or figures. |
|---|---|
| All unscheduled vi | isits will be included in listings. |
| Descriptive Summary | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 15.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to PKOne standards. Note: Concentration values will be imputed as per GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created. Dataset specification will be detailed in a separate document. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by Clinical Pharmacology Modelling and Simulation function will be created. Dataset specification will be detailed in a separate document. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: None |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to SOP_314000. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to PKOne. |

## 15.6. Appendix 6: Derived and Transformed Data

#### 15.6.1. General (Parts A and B)

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Dose Date → Study Day = Ref Date Dose Date</li>
  - Ref Data ≥ Dose Date → Study Day = Ref Date Dose Date + 1

## 15.6.2. Study Population

#### Age

- Only year of birth will be collected on the CRF and birth date will be presented in listings as 'YYYY'.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as '30<sup>th</sup>
  June' and then calculated based on the dose date.

## 15.6.3. Safety

#### **ECG Parameters**

#### RR Interval

- If RR interval (msec) is not provided directly, then RR can be derived as:
  - o If QTcF is machine read, then:

$$RR - \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value, then do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### Laboratory parameters

 If a laboratory value which is expected to have a numeric value for summary purposes, has a nondetectable level reported in the database, where the numeric value is missing, but typically a character

#### **ECG Parameters**

value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

- Example 1: 2 Significant Digits  $\rightarrow$  '< x' becomes x 0.01
- Example 2: 1 Significant Digit  $\rightarrow$  '> x' becomes x + 0.1
- Example 3: 0 Significant Digits  $\rightarrow$  '< x' becomes x 1

# 15.7. Appendix 7: Reporting Standards for Missing Data

## 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>In both Parts A and B, participant study completion (i.e. as specified in the protocol) is defined as having completed all phases of the study including the last scheduled assessment shown in the SoA (Section 15.2).</li> <li>Withdrawn participants may be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Section 15.3 or will be summarised as withdrawal visits. |

## 15.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated using a "blank" in participant listing displays, unless all data for a specific visit are missing (in which case the data is excluded from the table).</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |

## 15.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>In case of partial dates (i.e. day missing, only month and year present) recorded for AE start and end, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered Treatment Emergent as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the last contact date will be used.</li> </ul> </li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date: '01' will be used for the day if the month is not missing, and '01-Jan' will be used if both month and day are missing.</li> <li>If the partial date is a stop date: '28/29/30/31' will be used for the day if the month is not missing, and '31-Dec' will be used if both month and day are missing.</li> <li>For medications recorded in the eCRF as prior medications, the earlier of this imputed date or the day before the treatment start date will be used.</li> </ul> |

| Element | Reporting Detail |
|---------|----------------------------------------------------------|
| | The recorded partial date will be displayed in listings. |

# 15.8. Appendix 8: Values of Potential Clinical Importance

## 15.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (> x) |
| Haematocrit | Ratio of | Male | | 0.54 |
| Tidematociit | 1 | $\Delta$ from BL | ↓ 0.075 | |
| Haamaglahin | g/L | Male | | 180 |
| Haemoglobin | | $\Delta$ from BL | ↓ 25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Eosinophil Count | x10 <sup>9</sup> / L | | | 1 |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (> x) |
| Blood urea nitrogen | mmol/L | | | 10.5 |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | μmol/L | $\Delta$ from BL | | ↑ 26 |
| eGFR | ml/min/1.<br>73m <sup>2</sup> | | 60 | |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total Protein | g/L | | 50 | 85 |

| Liver Function | | | |
|--------------------|--------|----------|--------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2 x ULN |
| AST/SGOT | U/L | High | ≥ 2 x ULN |
| AlkPhos | U/L | High | ≥ 2 x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5 x ULN |
| | µmol/L | | ≥ 1.5 x ULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2 x ULN ALT |

## 15.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 15.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Temperature | °C | <35 | ≥37.5 |

# 15.8.4. Urinalysis

| Urinalysis | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| Bilirubin | | High | >1+ |
| Glucose | | High | >1+ |
| Ketone | | High | >2+ |
| Leukocytes (dipstick) | | High | >1+ |
| Nitrite | | High | Positive |
| Occult blood (dipstick) | | High | >1+ |
| ьЦ | | Low | <4.6 |
| pH | | High | >8 |
| Protein | | High | >1+ |
| RBC (microscopy) | cells/hpf | High | >3 |
| Chaoifia arouity | | Low | <1.001 |
| Specific gravity | | High | >1.035 |
| Urobilinogen | mg/dL | High | >1 |
| WBC (microscopy) | cells/hpf | High | >5 |

## 15.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

#### 15.9.1. Population Pharmacokinetic (PopPK) Dataset Specification

PopPK dataset specification will be provided as a separate document.

## 15.9.2. Population Pharmacokinetic (PopPK) Methodology

An exploratory graphical analysis of the drug plasma concentration-time data will be performed by generating the plots as presented in Appendix 12: List of Data Displays.

A previous PopPK model developed from the first time in human study 200630 (GSK Document Number 2017N352860\_00), incorporating linear and non-linear (target mediated drug disposition (TMDD), Michaelis-Menten) elimination pathways, will be used to fit the drug plasma concentration-time data. The model will be updated accordingly to describe the absorption profiles after SC doses of GSK2831781. For this update it will be assumed that the distribution and elimination of GSK2831781 will be the same regardless of the route of administration (IV or SC).

The appropriateness of the updated model will be assessed by the objective function value (OFV), successful convergence, covariance estimation, shrinkage, parameter uncertainty, standard Goodness-of-Fit (GoF) and simulation-based diagnostic plots e.g. Visual Predictive Check (VPC).

The GoF plots may include, but are not limited to:

- Population and individual predictions versus observations
- Conditional weighted residuals versus population predictions and time

If a VPC is done, this will be based on 1000 simulations with the model and the design structure of the observed data (i.e. dose level and time, time of PK sampling and individual values of model covariates, if any). The median and the 10th and 90th will be compared to the observed data. Stratification by dose level and administration route of GSK2831781 or geographic ancestry will be used.

The individual PK parameters will be computed from the PopPK model and will be summarised by treatment group and geographic ancestry.

# 15.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

#### 15.10.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

PK/PD dataset specification will be provided as a separate document.

#### 15.10.2. Pharmacokinetic / Pharmacodynamic Methodology

An exploratory graphical analysis of the drug effect on LAG3<sup>+</sup> cell depletion, sLAG3 concentrations and regulatory T cells count will be performed by generating the PD plots as presented in Appendix 12: List of Data Displays.

A previous indirect response model developed from all available cell depletion data from the first-time in human study 200630 (GSK Document Number 2017N352860\_00) will be fitted to the current PD data using the nonlinear mixed effects modelling software NONMEM. Data relative to CD4<sup>+</sup>CD45RA<sup>-</sup>1B4<sup>+</sup> cell count will be used to model T cell depletion.

The appropriateness of the PopPK/PD model will be assessed by the OFV, successful convergence, covariance estimation, shrinkage, parameter uncertainty, standard GoF and simulation-based diagnostic plots e.g. VPC.

The GoF plots may include, but are not limited to:

- Population and individual predictions versus observations
- Conditional weighted residuals versus population predictions and time

If a VPC is done, this will be based on 1000 simulations with the model and the design structure of the observed data (i.e. dose level and time, time of PD sampling and individual values of model covariates, if any). The median and the 10th and 90th will be compared to the observed data. Stratification by dose level and administration route of GSK2831781 or geographic ancestry will be used.

# 15.11. Appendix 11: Abbreviations & Trade Marks

## 15.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADA | Anti-drug antibody |
| AE | Adverse Event |
| ALT | Alanine aminotransaminase |
| ANOVA | Analysis of variance |
| AST | Aspartate Aminotransferase |
| AUC(0-t) | Area under the plasma concentration-time curve from time zero (pre-dose) to |
| , , | last time of quantifiable concentration |
| A&R | Analysis and Reporting |
| BUN | Blood Urea Nitrogen |
| CI | Confidence Interval |
| Cmax | Maximum observed plasma concentration |
| CMV | Cytomegalovirus |
| CPEM | Clinical Pharmacology and Experimental Medicine |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRF | Case Record Form |
| CSV | Comma-separated values |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| EBV | Epstein-Barr Virus |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| F | Bioavailability |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GCDO | Global Clinical & Data Operations |
| GCSD | Global Clinical Sciences & Delivery |
| GoF | Goodness-of-Fit |
| GSK | GlaxoSmithKline |
| HARP | Harmonized Analysis and Reporting Process |
| HbcAb | Hepatitis B core antibody |
| HbsAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| HIV | Human Immunodeficiency Virus |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| INR | International normalized ratio |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| IP. | Investigational Product |
| IV | Intravenous |
| LAG3 | Lymphocyte Activation Gene-3 |
| MCH | Mean Corpuscular Hemoglobin |
| MCV | Mean Corpuscular Volume |
| NQ | Non-quantifiable |
| OFV | Objective Function Value |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PKPD | Pharmacokinetic / Pharmacodynamic |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RBC | Red Blood Cell |
| RC | (Interim) Review Committee |
| RTF | Rich Text Format |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SGOT | Serum Glutamic-Oxaloacetic Transaminase |
| SGPT | Serum Glutamic-Pyruvic Transaminase |
| sLAG3 | Soluble LAG3 |
| SMG | Safety and Medical Governance |
| SoA | Schedule of Activities |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TB | Tuberculosis |
| TLF | Tables, Listings & Figures |
| tmax | Time of occurrence of Cmax |
| TMDD | Target Mediated Drug Disposition |
| ULN | Upper limit of normal |
| VPC | Visual Predictive Check |
| VZV | Varicella zoster virus |
| WBC | White Blood Cell |
| WNL | Windows Non-Linear |

## 15.11.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

None

# Trademarks not owned by the GlaxoSmithKline Group of Companies

NONMEM

SAS

WinNonlin

## 15.12. Appendix 12: List of Data Displays

## 15.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|-------------|
| Study Population | 1.1 to 1.20 | - |
| Safety | 2.1 to 2.34 | 2.1 to 2.2 |
| Pharmacokinetic | 3.1 to 3.8 | 3.1 to 3.4 |
| Population Pharmacokinetic (PopPK) | 4.1 to 4.x* | 4.1 to 4.x* |
| Pharmacodynamic | 5.1 to 5.7 | 5.1 to 5.10 |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.x* | 6.1 to 6.x* |
| Section | Listi | ngs |
| ICH Listings | 1 to 66 | |
| Other Listings | 67 to | ) X* |

<sup>\*</sup> PopPK and PK/PD displays will be generated by CPMS as needed; the number of displays is not predefined.

## 15.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|-------|---------|
| Study Population | - | - | POP_Ln |
| Safety | SAFE_Fn | - | SAFE_Ln |
| Pharmacokinetic | - | PK_Tn | - |
| Population Pharmacokinetic (PopPK) | - | - | - |
| Pharmacodynamic | PD_Fn | - | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | - | - | - |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 15.12.3. Deliverables

| Delivery | Description |
|----------|------------------------------------------------|
| IA | Interim Analysis Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |

# 15.12.4. Study Population Tables

## Part A

| Study I | Population Tab | les (Part A) | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Part A: Summary of Subject Disposition for the Subject Conclusion Record | Add footnote: Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK display standards. By treatment and geographic ancestry. | IA<br>SAC |
| 1.2. | Screened | ES6 | Part A: Summary of Screening Status and Reasons for Screen Failure | | SAC |
| Protoc | ol Deviation | | | | |
| 1.3. | Safety | DV1 | Part A: Summary of Important Protocol Deviations | By treatment and geographic ancestry. Include Total column. | SAC |
| Popula | tion Analysed | | | | |
| 1.4. | Screened | SP1 | Part A: Summary of Study Populations | By treatment and geographic ancestry. | IA<br>SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.5. | Safety | DM1 | Part A: Summary of Demographic Characteristics | By treatment and geographic ancestry. | IA<br>SAC |
| 1.6. | Safety | DM5 | Part A: Summary of Race and Racial Combinations | Only include race detail categories with >0 subjects. By treatment. | SAC |
| 1.7. | Randomized | DM11 | Part A: Summary of Age Ranges | By treatment and geographic ancestry. | SAC |
| Medica | I Conditions | | | | |

| Study F | Study Population Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Safety | MH1 | Part A: Summary of Past Medical Conditions | By treatment and geographic ancestry. | SAC |
| 1.9. | Safety | MH1 | Part A: Summary of Current Medical Conditions | By treatment and geographic ancestry. | SAC |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.10. | Safety | EX1 | Part A: Summary of Exposure to Study Treatment | By treatment and geographic ancestry. | SAC |

## Part B

| Study F | Population Tabl | les (Part B) | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.11. | Safety | ES1 | Part B: Summary of Subject Disposition for the Subject Conclusion Record | By treatment. | SAC |
| 1.12. | Screened | ES6 | Part B: Summary of Screening Status and Reasons for Screen Failure | | SAC |
| Protoco | ol Deviation | | | | |
| 1.13. | Safety | DV1 | Part B: Summary of Important Protocol Deviations | By treatment. Include Total column. | SAC |
| Popula | Population Analysed | | | | |
| 1.14. | Screened | SP1 | Part B: Summary of Study Populations | By treatment. | SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.15. | Safety | DM1 | Part B: Summary of Demographic Characteristics | By treatment. | SAC |

| Study F | Study Population Tables (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.16. | Safety | DM5 | Part B: Summary of Race and Racial Combinations | Only include race detail categories with >0 subjects. By treatment. | SAC |
| 1.17. | Randomized | DM11 | Part B: Summary of Age Ranges | By treatment. | SAC |
| Medica | Conditions | | | | |
| 1.18. | Safety | MH1 | Part B: Summary of Past Medical Conditions | By treatment. | SAC |
| 1.19. | Safety | MH1 | Part B: Summary of Current Medical Conditions | By treatment. | SAC |
| Exposu | exposure and Treatment Compliance | | | | |
| 1.20. | Safety | EX1 | Part B: Summary of Exposure to Study Treatment | By treatment. | SAC |

# 15.12.5. Safety Tables

## Part A

| Safety | Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Part A: Summary of All Adverse Events by System Organ Class and Preferred Term | IA: By geographic ancestry. SAC: By treatment and geographic ancestry. | IA<br>SAC |
| 2.2. | Safety | AE3 | Part A: Summary of Drug-Related Adverse Events | IA: By geographic ancestry. SAC: By treatment and geographic ancestry. | IA<br>SAC |
| 2.3. | Safety | AE3 | Part A: Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency | By treatment and geographic ancestry. | SAC |
| 2.4. | Safety | AE5A | Part A: Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | Page by treatment and geographic ancestry. | SAC |
| 2.5. | Safety | AE5A | Part A: Summary of Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | Page by treatment and geographic ancestry. | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 2.6. | Safety | AE16 | Part A: Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | IA: By geographic ancestry. SAC: By treatment and geographic ancestry. | IA<br>SAC |
| 2.7. | Safety | AE3 | Part A: Summary of Serious Drug-Related Adverse Events by Overall Frequency | IA: By geographic ancestry. SAC: By treatment and geographic ancestry. | IA<br>SAC |
| 2.8. | Safety | AE3 | Part A: Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | By treatment and geographic ancestry. | SAC |

| Safety | Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Chemistry | / | | | |
| 2.9. | Safety | LB1 | Part A: Summary of Chemistry Changes from Baseline | By treatment and geographic ancestry. | SAC |
| Labora | tory: Haematol | ogy | | | |
| 2.10. | Safety | LB1 | Part A: Summary of Haematology Changes from Baseline | By treatment and geographic ancestry. IA: Only include the following parameters: Neutrophils, Lymphocytes. | IA<br>SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | |
| 2.11. | Safety | LB1 | Part A: Summary of Urine Concentration Changes from Baseline | By treatment and geographic ancestry. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.12. | Safety | LIVER1 | Part A: Summary of Liver Monitoring/Stopping Event Reporting | By treatment and geographic ancestry. | IA<br>SAC |
| 2.13. | Safety | LIVER10 | Part A: Summary of Hepatobiliary Laboratory Abnormalities | By treatment and geographic ancestry. | SAC |
| ECG | 1 | | | | |
| 2.14. | Safety | EG1 | Part A: Summary of ECG Findings | By treatment and geographic ancestry. | SAC |
| 2.15. | Safety | EG10 | Part A: Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | By treatment and geographic ancestry. | SAC |
| 2.16. | Safety | EG2 | Part A: Summary of Change from Baseline in ECG Values by Visit | By treatment and geographic ancestry. | SAC |
| Vital Si | gns | | | | |
| 2.17. | Safety | VS1 | Part A: Summary of Change from Baseline in Vital Signs | By treatment and geographic ancestry. | SAC |

## Part B

| Safety | Safety Tables (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | dverse Events (AEs) | | | | |
| 2.18. | Safety | AE1 | Part B: Summary of All Adverse Events by System Organ Class and Preferred Term | By treatment. | SAC |
| 2.19. | Safety | AE3 | Part B: Summary of Drug-Related Adverse Events | By treatment. | SAC |
| 2.20. | Safety | AE3 | Part B: Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency | By treatment. | SAC |
| 2.21. | Safety | AE5A | Part B: Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | Page by treatment. | SAC |
| 2.22. | Safety | AE5A | Part B: Summary of Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | Page by treatment. | SAC |
| Serious | and Other Sig | nificant Adverse I | | | |
| 2.23. | Safety | AE16 | Part B: Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | By treatment. | SAC |
| 2.24. | Safety | AE3 | Part B: Summary of Serious Drug-Related Adverse Events by Overall Frequency | By treatment. | SAC |
| 2.25. | Safety | AE3 | Part B: Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | By treatment. | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 2.26. | Safety | LB1 | Part B: Summary of Chemistry Changes from Baseline | By treatment. | SAC |
| Labora | tory: Haematol | ogy | | | |
| 2.27. | Safety | LB1 | Part B: Summary of Haematology Changes from Baseline | By treatment. | SAC |

| Safety | Tables (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | <b>5</b> | | | |
| 2.28. | Safety | LB1 | Part B: Summary of Urine Concentration Changes from Baseline | By treatment. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.29. | Safety | LIVER1 | Part B: Summary of Liver Monitoring/Stopping Event Reporting | By treatment. | SAC |
| 2.30. | Safety | LIVER10 | Part B: Summary of Hepatobiliary Laboratory Abnormalities | By treatment. | SAC |
| ECG | | | | | |
| 2.31. | Safety | EG1 | Part B: Summary of ECG Findings | By treatment. | SAC |
| 2.32. | Safety | EG10 | Part B: Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | By treatment. | SAC |
| 2.33. | Safety | EG2 | Part B: Summary of Change from Baseline in ECG Values by Visit | By treatment. | SAC |
| Vital Si | gns | | | | - |
| 2.34. | Safety | VS1 | Part B: Summary of Change from Baseline in Vital Signs | By treatment. | SAC |

# 15.12.6. Safety Figures

## Part A

| Pharma | Pharmacokinetic Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Haematol | ogy | | | |
| 2.1. | Safety | [Non-standard]<br>SAFE_F1 | Part A: Individual Plots of Haematology | By treatment and geographic ancestry. Only include the following parameters: Neutrophils, Lymphocytes. | IA |
| 2.2. | Safety | [Non-standard]<br>SAFE_F2 | Part A: Mean (±SD) Plots of Haematology | By treatment and geographic ancestry. Only include the following parameters: Neutrophils, Lymphocytes. | IA |

## 15.12.7. Pharmacokinetic Tables

## Part A

| Pharma | Pharmacokinetic Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic Con | centrations | | | |
| 3.1. | PK | PK01 | Part A: Summary of GSK2831781 Plasma Pharmacokinetic Concentration-Time Data | Include 95% Confidence Interval for the mean. By treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |
| Pharma | cokinetic Para | meters | | | |
| 3.2. | PK | PK03 | Part A: Summary of Derived GSK2831781 Plasma<br>Pharmacokinetic Parameters | Include 95% Confidence Interval for the mean. By treatment and geographic ancestry. | IA<br>SAC |
| 3.3. | PK | PK05 | Part A: Summary of Log-Transformed Derived GSK2831781 Plasma Pharmacokinetic Parameters | By treatment and geographic ancestry. | IA<br>SAC |
| Pharma | Pharmacokinetic Statistical Analyses | | | | |
| 3.4. | PK | [Non-standard]<br>PK_T1 | Part A: Table of Ethnosensitivity Model Results | | SAC |

## Part B

| Pharma | Pharmacokinetic Tables (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic Con | centrations | | | |
| 3.5. | PK | PK01 | Part B: Summary of GSK2831781 Plasma Pharmacokinetic Concentration-Time Data | Include 95% Confidence Interval for the mean. By treatment. | SAC |
| Pharma | cokinetic Para | meters | | | |
| 3.6. | PK | PK03 | Part B: Summary of Derived GSK2831781 Plasma<br>Pharmacokinetic Parameters | Include 95% Confidence Interval for the mean. By treatment. | SAC |
| 3.7. | PK | PK05 | Part B: Summary of Log-Transformed Derived GSK2831781 Plasma Pharmacokinetic Parameters | By treatment. | SAC |
| Pharma | Pharmacokinetic Statistical Analyses | | | | |
| 3.8. | PK | [Non-standard]<br>PK_T1 | Part B: Table of Bioavailability Model Results | | SAC |

# 15.12.8. Pharmacokinetic Figures

## Part A

| Pharma | Pharmacokinetic Figures (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic Con | centrations | | | |
| 3.1. | PK | PK24 | Part A: Individual GSK2831781 Plasma Concentration-Time Plots (Linear and Semi-log) by Treatment and Geographic Ancestry | By treatment and geographic ancestry. IA: do not show subject IDs. Different colours and symbols for treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |
| 3.2. | PK | PK19 | Part A: Mean (±SD) GSK2831781 Plasma Concentration-Time Plots (Linear and Semi-log) by Treatment and Geographic Ancestry | By treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |

## Part B

| Pharmacokinetic Figures (Part B) | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic Cond | centrations | | | |
| 3.3. | PK | PK24 | Part B: Individual GSK2831781 Plasma Concentration-Time Plots (Linear and Semi-log) by Treatment | By treatment. | SAC |
| 3.4. | PK | PK19 | Part B: Mean (±SD) GSK2831781 Plasma Concentration-Time Plots (Linear and Semi-log) by Treatment | By treatment. | SAC |

# 15.12.9. Pharmacokinetic Population (PopPK) Tables

Tables will be generated by CPMS as needed for part A & B.

# 15.12.10. Pharmacokinetic Population (PopPK) Figures

Figures will be generated by CPMS as needed for part A & B.

# 15.12.11. Pharmacodynamic Tables

## Part A

| Pharma | Pharmacodynamic Tables (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| LAG3+ | T Cells | | | | |
| 5.1. | Safety | PD1 | Part A: Summary of LAG3+ T Cells in Blood by Visit | Absolute, %CFB. By treatment and geographic ancestry. By cell populations as defined in 11.1.1. IA: only include data up to Day 29. | IA<br>SAC |
| Soluble | LAG3 | | | | |
| 5.2. | Safety | PD1 | Part A: Summary of sLAG3 in Blood by Visit | Absolute, %CFB. By treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |
| Regulat | tory T Cells | | | | |
| 5.3. | Safety | PD1 | Part A: Summary of Regulatory T Cells in Blood by Visit | Absolute, %CFB. By treatment. | SAC |
| Immuno | ogenicity | | | | |
| 5.4. | Safety | IMM1 | Part A: Summary of Positive Immunogenicity Results | | SAC |

## Part B

| Pharma | Pharmacodynamic Tables (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| LAG3+ | T Cells | | | | |
| 5.5. | Safety | PD1 | Part B: Summary of LAG3+ T Cells in Blood by Visit | Absolute, %CFB. By treatment. By cell populations as defined in 11.1.1. | SAC |
| Soluble | LAG3 | | | | |
| 5.6. | Safety | PD1 | Part B: Summary of sLAG3 in Blood by Visit | Absolute, %CFB. By treatment. | SAC |
| Immun | mmunogenicity | | | | |
| 5.7. | Safety | IMM1 | Part B: Summary of Positive Immunogenicity Results | | SAC |

# 15.12.12. Pharmacodynamic Figures

## Part A

| Pharma | Pharmacodynamic Figures (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| LAG3+ | LAG3+ T Cells | | | | |
| 5.1. | Safety | [Non-standard]<br>PD_F1 | Part A: Individual Plot of LAG3+ T Cells in Blood Over Time | Absolute, %CFB. By treatment and geographic ancestry. Page by cell population, as defined in 11.1.1. IA: do not show subject IDs. Different colours and symbols for treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |
| 5.2. | Safety | [Non-standard]<br>PD_F2 | Part A: Mean (±SD) Plot of LAG3+ T Cells in Blood Over Time | Absolute, %CFB. By treatment and geographic ancestry. Page by cell population, as defined in 11.1.1. IA: only include data up to Day 29. | IA<br>SAC |
| Soluble | LAG3 | | | | |
| 5.3. | Safety | [Non-standard]<br>PD_F1 | Part A: Individual Plot of sLAG3 in Blood Over Time | Absolute, %CFB. By treatment and geographic ancestry. IA: do not show subject IDs. Different colours and symbols for treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |
| 5.4. | Safety | [Non-standard]<br>PD_F2 | Part A: Mean (±SD) Plot of sLAG3 in Blood Over Time | Absolute, %CFB. By treatment and geographic ancestry. IA: only include data up to Day 29. | IA<br>SAC |

| Regulat | Regulatory T Cells | | | | |
|---|---|---|---|---|---|
| 5.5. | Safety | [Non-standard]<br>PD_F1 | Part A: Individual Plot of Regulatory T Cells in Blood Over Time | Absolute, %CFB. By treatment. | SAC |
| 5.6. | Safety | [Non-standard]<br>PD_F2 | Part A: Mean (±SD) Plot of Regulatory T Cells in Blood Over Time | Absolute, %CFB. By treatment. | SAC |

## Part B

| Pharma | Pharmacodynamic Figures (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| LAG3+ | T Cells | | | | |
| 5.7. | Safety | [Non-standard]<br>PD_F1 | Part B: Individual Plot of LAG3+ T Cells in Blood Over Time | Absolute, %CFB. By treatment. Page by cell population, as defined in 11.1.1. | SAC |
| 5.8. | Safety | [Non-standard]<br>PD_F2 | Part B: Mean (±SD) Plot of LAG3+ T Cells in Blood Over Time | Absolute, %CFB. By treatment. Page by cell population, as defined in 11.1.1. | SAC |
| Soluble | LAG3 | | | | |
| 5.9. | Safety | [Non-standard]<br>PD_F1 | Part B: Individual Plot of sLAG3 in Blood Over Time | Absolute, %CFB. By treatment. | SAC |
| 5.10. | Safety | [Non-standard]<br>PD_F2 | Part B: Mean (±SD) Plot of sLAG3 in Blood Over Time | Absolute, %CFB. By treatment. | SAC |

# 15.12.13. Pharmacokinetic / Pharmacodynamic Tables

Tables will be generated by CPMS as needed for part A & B.

# 15.12.14. Pharmacokinetic / Pharmacodynamic Figures

Figures will be generated by CPMS as needed for part A & B.

# 15.12.15. ICH Listings

## Part A

| ICH Lis | stings (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Safety | ES2 | Part A: Listing of Reasons for Study Withdrawal | | SAC |
| 2. | Screened | ES7 | Part A: Listing of Reasons for Screen Failure | | SAC |
| 3. | Safety | SD2 | Part A: Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 4. | Safety | BL1 | Part A: Listing of Subjects for Whom the Treatment Blind was Broken | | SAC |
| 5. | Safety | TA1 | Part A: Listing of Planned and Actual Treatments | | SAC |
| Protoc | ol Deviations | | | | • |
| 6. | Safety | DV2 | Part A: Listing of Important Protocol Deviations | | SAC |
| 7. | Safety | IE3 | Part A: Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | ations Analysed | | | | |
| 8. | Screened | SP3 | Part A: Listing of Subjects Excluded from Any Population | | SAC |
| Demog | graphic and Baseli | ine Characteristics | | | • |
| 9. | Safety | DM2 | Part A: Listing of Demographic Characteristics | | SAC |
| 10. | Safety | DM9 | Part A: Listing of Race | | SAC |
| Medica | al Conditions and | Prior/Concomitant I | Medications | | |
| 11. | Safety | MH2 | Part A: Listing of Current/Past Medical Conditions | | SAC |
| 12. | Safety | CM2 | Part A: Listing of Concomitant Medications | | SAC |

| ICH Li | stings (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | ure and Treatmen | t Compliance | | | • |
| 13. | Safety | EX3 | Part A: Listing of Exposure Data | | SAC |
| Adver | se Events | | | | |
| 14. | Safety | AE7 | Part A: Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 15. | Safety | AE8 | Part A: Listing of All Adverse Events | | IA<br>SAC |
| 16. | Safety | AE2 | Part A: Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Seriou | s and Other Signi | ficant Adverse Even | ts | | • |
| 17. | Safety | AE8CPA | Part A: Listing of Serious Adverse Events (Fatal & Non-Fatal) | Include fatal and non-fatal status | SAC |
| 18. | Safety | AE8 | Part A: Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | SAC |
| 19. | Safety | AE8 | Part A: Listing of Other Significant Adverse Events | | SAC |
| 20. | Safety | AE14 | Part A: Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| Hepat | obiliary (Liver) | | | | • |
| 21. | Safety | MH2 | Part A: Listing of Medical Conditions for Subjects with Liver Stopping Events | | SAC |
| 22. | Safety | SU2 | Part A: Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| 23. | Safety | LIVER6 | Part A: Listing of Liver Stopping Event Information for RUCAM Score | | SAC |
| 24. | Safety | LIVER7 | Part A: Listing of Liver Biopsy Details | | SAC |

| ICH Lis | stings (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 25. | Safety | LIVER8 | Part A: Listing of Liver Imaging Details | | SAC |
| All Lab | oratory | | | | |
| 26. | Safety | LB5 | Part A: Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 27. | Safety | LB5 | Part A: Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 28. | Safety | LB14 | Part A: Listing of Laboratory Data with Character Results | IA: Only include the following parameters: Neutrophils, Lymphocytes | IA<br>SAC |
| 29. | Safety | UR2A | Part A: Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| ECG | | | | | |
| 30. | Safety | EG3 | Part A: Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 31. | Safety | EG3 | Part A: Listing of ECG Values of Potential Clinical Importance | | SAC |
| 32. | Safety | EG5 | Part A: Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | | SAC |
| Vital S | igns | | | | |
| 33. | Safety | VS4 | Part A: Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

## Part B

| ICH Lis | stings (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | · |
| 34. | Safety | ES2 | Part B: Listing of Reasons for Study Withdrawal | | SAC |
| 35. | Screened | ES7 | Part B: Listing of Reasons for Screen Failure | | SAC |
| 36. | Safety | SD2 | Part B: Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 37. | Safety | BL1 | Part B: Listing of Subjects for Whom the Treatment Blind was Broken | | SAC |
| 38. | Safety | TA1 | Part B: Listing of Planned and Actual Treatments | | SAC |
| Protoc | ol Deviations | | | | |
| 39. | Safety | DV2 | Part B: Listing of Important Protocol Deviations | | SAC |
| 40. | Safety | IE3 | Part B: Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 41. | Screened | SP3 | Part B: Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 42. | Safety | DM2 | Part B: Listing of Demographic Characteristics | | SAC |
| 43. | Safety | DM9 | Part B: Listing of Race | | SAC |
| Medica | I Conditions ar | nd Prior/Concomit | ant Medications | | · |
| 44. | Safety | MH2 | Part B: Listing of Current/Past Medical Conditions | | SAC |
| 45. | Safety | CM2 | Part B: Listing of Concomitant Medications | | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 46. | Safety | EX3 | Part B: Listing of Exposure Data | | SAC |

| ICH Lis | tings (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | • |
| 47. | Safety | AE7 | Part B: Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 48. | Safety | AE8 | Part B: Listing of All Adverse Events | | SAC |
| 49. | Safety | AE2 | Part B: Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious | and Other Sig | nificant Adverse l | Events | | |
| 50. | Safety | AE8CPA | Part B: Listing of Serious Adverse Events (Fatal & Non-Fatal) | Include fatal and non-fatal status | SAC |
| 51. | Safety | AE8 | Part B: Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | SAC |
| 52. | Safety | AE8 | Part B: Listing of Other Significant Adverse Events | | SAC |
| 53. | Safety | AE14 | Part B: Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| Hepato | biliary (Liver) | | | , | |
| 54. | Safety | MH2 | Part B: Listing of Medical Conditions for Subjects with Liver Stopping Events | | SAC |
| 55. | Safety | SU2 | Part B: Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| 56. | Safety | LIVER6 | Part B: Listing of Liver Stopping Event Information for RUCAM Score | | SAC |
| 57. | Safety | LIVER7 | Part B: Listing of Liver Biopsy Details | | SAC |
| 58. | Safety | LIVER8 | Part B: Listing of Liver Imaging Details | | SAC |
| All Lab | oratory | | | | |
| 59. | Safety | LB5 | Part B: Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | SAC |

| ICH Lis | ICH Listings (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 60. | Safety | LB5 | Part B: Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 61. | Safety | LB14 | Part B: Listing of Laboratory Data with Character Results | | SAC |
| 62. | Safety | UR2A | Part B: Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| ECG | | | | | |
| 63. | Safety | EG3 | Part B: Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 64. | Safety | EG3 | Part B: Listing of ECG Values of Potential Clinical Importance | | SAC |
| 65. | Safety | EG5 | Part B: Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | | SAC |
| Vital Si | Vital Signs | | | | |
| 66. | Safety | VS4 | Part B: Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

# 15.12.16. Non-ICH Listings

# Part A

| Non-IC | Non-ICH Listings (Part A) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 67. | Safety | [Non-standard]<br>POP_L1 | Part A: Listing of Dose Dispensation Deviations | By geographic ancestry. | IA |
| Pharma | acokinetic Data | | | | |
| 68. | PK | PK07 | Part A: Listing of GSK2831781 Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 69. | PK | PK13 | Part A: Listing of Derived GSK2831781 Plasma Pharmacokinetic Parameters | | SAC |
| Pharma | acodynamic: L/ | AG3+ T Cells | | | |
| 70. | Safety | [Non-standard]<br>PD_L1 | Part A: Listing of LAG3+ T cells in Blood | | SAC |
| Pharma | acodynamic: So | oluble LAG3 | | | |
| 71. | Safety | [Non-standard]<br>PD_L1 | Part A: Listing of sLAG3 in Blood | | SAC |
| Pharma | acodynamic: Ro | egulatory T Cells | | | |
| 72. | Safety | [Non-standard]<br>PD_L1 | Part A: Listing of Regulatory T Cells in Blood | | SAC |
| Pharma | acodynamic: Im | nmunogenicity | | | |
| 73. | Safety | IMM2 | Part A: Listing of Immunogenicity Results | | SAC |

## Part B

| Non-ICI | Non-ICH Listings (Part B) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Local T | olerability | | | | |
| 74. | Safety | [Non-standard]<br>SAFE_L1 | Part B: Listing of Injection Sites and Injection Site Reactions | | SAC |
| Pharma | cokinetic Data | | | | |
| 75. | PK | PK07 | Part B: Listing of GSK2831781 Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 76. | PK | PK13 | Part B: Listing of Derived GSK2831781 Plasma Pharmacokinetic Parameters | | SAC |
| Pharma | codynamic: LA | AG3+ T Cells | | | |
| 77. | Safety | [Non-standard]<br>PD_L1 | Part B: Listing of LAG3+ T Cells in Blood | | SAC |
| Pharma | codynamic: So | oluble LAG3 | | | |
| 78. | Safety | [Non-standard]<br>PD_L1 | Part B: Listing of sLAG3 in Blood | | SAC |
| Pharma | Pharmacodynamic: Immunogenicity | | | | |
| 79. | Safety | IMM2 | Part B: Listing of Immunogenicity Results | | SAC |

# 15.13. Appendix 13: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request